CLINICAL TRIAL: NCT02961582
Title: Effectiveness and Cost-effectiveness of Sacral Neuromodulation in Patients With Idiopathic Slow-transit Constipation Refractory to Conservative Treatments
Brief Title: Effectiveness and Cost-effectiveness of Sacral Neuromodulation in Patients With Idiopathic Slow-transit Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch National Health Care Institute (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL57367.068.16
Record Dates: First submitted 2016-10-12; First posted 2016-11-11 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Constipation; Surgery
Keywords: Sacral neuromodulation; Constipation; Slow-transit constipation; Surgery; Colorectal surgery; Cost-effectiveness; Quality of life
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacral Neuromodulation (Experimental)
  Interventions: Device: Sacral Neuromodulation
- Personalized Conservative Treatment (Other)
  Interventions: Other: Personalized Conservative Treatment

INTERVENTIONS:
Device: Sacral Neuromodulation — SNM starts with a screening phase. In this phase a tined lead is inserted into the third sacral foramen and attached to an external stimulator, after which the patient enters a four-week stimulation test period. If the screening phase is successful (defecation frequency (DF) ≥3 a week), the external stimulator is changed for a pacemaker that is implanted in the buttocks. If the screening phase is unsuccessful (DF <3 a week), the lead is explanted.
  Patients in the intervention group are asked to limit the use of additional conservative treatments for constipation (such as laxatives and colonic irrigation) to what is necessary to relieve (the most severe) complaints. What is necessary to relieve complaints is determined by the patient.
  Other Names: Medtronic Interstim Therapy System
  Arms: Sacral Neuromodulation
Other: Personalized Conservative Treatment — The control group will receive the best and least invasive alternative treatment, which is personalized conservative treatment (PCT). PCT includes, a combination of laxative/medication use and/or colonic irrigation, depending on the preferences of the patient. Use of PCT will be documented.
  Other Names: Care as usual
  Arms: Personalized Conservative Treatment

SUMMARY:
Rationale: Previous reviews showed that the evidence regarding the effectiveness of sacral neuromodulation (SNM) in patients with therapy-resistant, idiopathic (slow-transit) constipation is of suboptimal quality. Furthermore, there is no estimate of costs and cost-effectiveness in this patient group.

Objective: The main objective of this study is to assess the effectiveness of SNM compared to personalized conservative treatment (PCT), in patients with idiopathic slow-transit constipation who are refractory to conservative treatment. The secondary objectives are assessing the 1) costs, 2) cost-effectiveness and 3) budget-impact of SNM compared to PCT.

Hypothesis: Based on previous research we hypothesize that SNM will be more effective than PCT in terms of a significantly higher proportion of patients having treatment success at 6 months.

Study design: An open-label pragmatic randomized controlled trial (RCT) combined with a prospective cohort study.

Study population: Adolescent (14-17 years) and adult (18-80 years) patients with idiopathic slow-transit constipation refractory to conservative treatment.

Intervention: The intervention is SNM, a minimally invasive surgical procedure consisting of two phases. In the screening phase an electrode is inserted near the third sacral nerve and connected to an external stimulator. If the screening phase is successful (average defecation frequency (DF) ≥3 a week), the electrode is connected to a pacemaker that is implanted in the buttocks of the patient. If not successful, patients receive conservative treatment. The control intervention is PCT. This is the best and least invasive alternative to SNM. PCT consists of medication and/or retrograde colonic irrigation.

Main study parameters/endpoints: The primary outcome is success at 6 months, defined as an average DF of ≥3 a week according to a 3-week defecation diary. Secondary outcomes are straining, sense of incomplete evacuation, constipation severity, fatigue, constipation specific and generic (health-related) quality of life ((HR)QOL), and costs at 6 months. Furthermore, cost-effectiveness and budget-impact will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* An average defecation frequency (DF) of <3 per week based on a 3-week defecation diary (patient-reported)
* Meet at least one other criterion of the Rome-IV criteria for idiopathic constipation based on the 3-week defecation diary (1)
* Refractory to conservative treatment
* Age: 14-80 years
* Slow-transit constipation

  (1) Rome-IV criteria for idiopathic constipation:
* Straining during ≥25% of defecations
* Lumpy or hard stools in ≥25% of defecations
* Sensation of incomplete evacuation for ≥25% of defecations
* Sensation of anorectal obstruction/blockage for ≥25% of defecations
* Manual manoeuvres to facilitate ≥25% of defecations

Exclusion Criteria:

* Obstructed outlet syndrome (objectified by defeacography)
* Irritable bowel syndrome (Rome-IV criteria for irritable bowel syndrome)
* Congenital or organic bowel pathology
* Rectal prolapse
* Anatomical limitations preventing placement of an electrode
* Skin and perineal disease with risk of infection
* Previous large bowel/rectal surgery
* Stoma
* Coexisting neurological disease
* Significant psychological co-morbidity as assessed subjectively by the investigator
* Being or attempting to become pregnant during study follow-up

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment success at 6 months | 6 months
  Treatment success is defined as an average defecation frequency of ≥ 3 a week based on a patient-reported defecation diary over a period of 3 weeks

SECONDARY OUTCOMES:
Defecation frequency | 1 and 3 months
  Defecation frequency based on a patient-reported defecation diary over a period of 3 weeks
Proportion of patients with a 50% reduction in the proportion of defecations with straining | Baseline, 1, 3 and 6 months
  The proportion of defecations with straining is derived from the data in the 3 week defecation diary. The reported proportion of defecations with straining is compared with the proportion of defecations with straining at baseline. Patients are divided in two groups: 1) ≥50% reduction in the proportion of defecations with straining and 2) <50% reduction in the proportion of defecations with straining.
Proportion of patients with a 50% reduction in the proportion of defecations with a sense of incomplete evacuation | Baseline, 1, 3 and 6 months
  The proportion of defecations with a sense of incomplete evacuation is derived from the data in the 3 week defecation diary. The reported proportion of defecations with a sense of incomplete evacuation is compared with the proportion of defecations with a sense of incomplete evacuation at baseline. Patients are divided in two groups: 1) ≥50% reduction in the proportion of defecations with a sense of incomplete evacuation and 2) <50% reduction in the proportion of defecations with a sense of incomplete evacuation.
Constipation severity | Baseline, 1, 3 and 6 months
  Displayed with the score from the Wexner constipation score (WCS).
Fatigue | Baseline, 1, 3 and 6 months
  Displayed with the score from the Fatigue Questionnaire (in Dutch 'Verkorte vermoeidheidsvragenlijst' (VVV)) .
Constipation-specific (health-related) quality of life ((HR)QOL) | Baseline, 1, 3 and 6 months
  Displayed with the score from the Patient Assessment of Constipation - Quality of Life (PAC-QOL) questionnaire
Generic (HR)QOL | Baseline, 1, 3 and 6 months
  In adults displayed with the score from the EQ-5D-5L and ICECAP-A In adolescents displayed with the score from the EQ-5D-5L and KIDSCREEN-27
Adverse events/complications | Baseline, 1, 3 and 6 months
  Reported by the clinician in a case report form (CRF)
Resource use/costs | Baseline, 3 and 6 months
  Health care costs, patient and family costs and costs outside the health care sector
Cost-effectiveness | 6 months
  Both from a societal and health care perspective, derived from the EQ-5D-5L scores and cost data obtained in this RCT
Budget-impact | 6 months
  From a societal, health care and health care insurance perspective, derived from the EQ-5D-5L scores and cost data obtained in this RCT

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie O Breukink, Dr., Principal Investigator — Maastricht University Medical Centre+; Carmen D Dirksen, Prof. dr., Principal Investigator — Maastricht University Medical Centre+
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Groene Hart Ziekenhuis, Gouda, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575
- [Background] Suares NC, Ford AC. Prevalence of, and risk factors for, chronic idiopathic constipation in the community: systematic review and meta-analysis. Am J Gastroenterol. 2011 Sep;106(9):1582-91; quiz 1581, 1592. doi: 10.1038/ajg.2011.164. Epub 2011 May 24. PMID 21606976
- [Background] van Wunnik BP, Peeters B, Govaert B, Nieman FH, Benninga MA, Baeten CG. Sacral neuromodulation therapy: a promising treatment for adolescents with refractory functional constipation. Dis Colon Rectum. 2012 Mar;55(3):278-85. doi: 10.1097/DCR.0b013e3182405c61. PMID 22469794
- [Background] Heemskerk SCM, Rotteveel AH, Benninga MA, Baeten CIM, Masclee AAM, Melenhorst J, van Kuijk SMJ, Dirksen CD, Breukink SO. Sacral neuromodulation versus personalized conservative treatment in patients with idiopathic slow-transit constipation: study protocol of the No.2-trial, a multicenter open-label randomized controlled trial and cost-effectiveness analysis. Int J Colorectal Dis. 2018 Apr;33(4):493-501. doi: 10.1007/s00384-018-2978-x. Epub 2018 Feb 22. PMID 29470731
- [Derived] Heemskerk SCM, Dirksen CD, van Kuijk SMJ, Benninga MA, Baeten CIM, Masclee AAM, Melenhorst J, Breukink SO. Sacral Neuromodulation Versus Conservative Treatment for Refractory Idiopathic Slow-transit Constipation: The Randomized Clinical No.2-Trial. Ann Surg. 2024 May 1;279(5):746-754. doi: 10.1097/SLA.0000000000006158. Epub 2023 Nov 23. PMID 37991178